CLINICAL TRIAL: NCT00017628
Title: Phase I Study of High-Dose Cyclophosphamide and Total Body Irradiation With T Lymphocyte-Depleted Autologous Peripheral Blood Stem Cell or Bone Marrow Rescue in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern Memorial Hospital (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/14975; NU-95MS1
Record Dates: First submitted 2001-06-06; First posted 2001-06-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Multiple Sclerosis; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Cyclophosphamide; Filgrastim; Methylprednisolone

INTERVENTIONS:
Drug: cyclophosphamide
Drug: filgrastim
Drug: methylprednisolone
Procedure: Autologous Stem Cell Transplantation

SUMMARY:
OBJECTIVES:

I. Determine the efficacy, in terms of disease progression, of high-dose cyclophosphamide and total body irradiation with T lymphocyte-depleted autologous peripheral blood stem cell or bone marrow rescue in patients with multiple sclerosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Following an induction course of cyclophosphamide IV, patients receive filgrastim (G-CSF) subcutaneously (SC) daily until the completion of peripheral blood stem cell (PBSC) harvesting. PBSCs are collected over several days. Patients who do not mobilize sufficient cells undergo bone marrow harvest. Harvested PBSCs or bone marrow then undergo T-lymphocyte depletion.

Patients receive cyclophosphamide IV over 1 hour on days -6 and -5 and methylprednisolone IV daily on days -4 to -1. Patients also undergo total body irradiation twice a day on days -4 to -1. Lymphocyte-depleted PBSCs or bone marrow is reinfused on day 0. Patients receive G-CSF SC daily beginning on day 0 and continuing until blood counts have recovered for 3 days.

Patients are followed at 1, 2, 3, 6, and 12 months and then annually for 5 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of multiple sclerosis Kurtzke score of 4.0-7.5 Increase of 1.0 point over the past 12 months More than 3 relapses in 24 months despite conventional disease modifying therapy Failure to stabilize active clinical progression with a 3-day regimen of methylprednisolone IV

--Prior/Concurrent Therapy--

Chemotherapy: No prior cladribine

Radiotherapy: No prior radiotherapy to greater than 10 cm2 of lung tissue No prior craniospinal irradiation No prior total lymphoid irradiation

--Patient Characteristics--

Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL

Hepatic: Hepatitis B antigen negative Bilirubin no greater than 2.0 mg/dL Transaminases no greater than 2 times upper limit of normal

Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No history of coronary artery disease Resting LVEF at least 45%

Pulmonary: FEV1/FVC at least 75% predicted DLCO at least 50% predicted

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No uncontrolled diabetes mellitus
* No other concurrent medical illness that would preclude study
* No concurrent psychiatric illness or mental deficiency that would preclude study
* No prior malignancy except localized basal cell or squamous cell skin cancer (malignancies judged to be cured by local surgical therapy such as head and neck cancer or stage I breast cancer, are considered on an individual basis)
* No presence of body shrapnel, metal fragments, or unremovable devices such as a pacemaker or aneurysm clip

Ages: 0 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Burt, Study Chair — Northwestern Memorial Hospital
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois